CLINICAL TRIAL: NCT07330661
Title: Neurointerdisciplinary Nursing Prevention Strategies for Deep Vein Thrombosis (DVT) After Neurosurgical Procedures: A Multicenter Randomized Controlled Trial and Nomogram Development
Brief Title: Nursing-Led Deep Vein Thrombosis Prevention in Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WestChinaH-HX-2025-010
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-12

CONDITIONS: Deep Vein Thrombosis (DVT)
Keywords: Neurosurgery; Interdisciplinary Nursing; Multimodal Prevention; Risk Prediction; Randomized Controlled Trial
MeSH Terms: conditions — Venous Thrombosis | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led prevention group (Experimental): In addition to routine post-operative care, participants assigned to the nurse-led prevention arm receive:
  * Graded early-movement plan starting within 24 h of surgery
  * Unconscious patients: passive leg exercises 10-15 min, 3× daily
  * Conscious patients: assisted leg, sitting and walking sessions escalated daily (target ≥ 40 min total activity, logged automatically by a wrist-band activity tracker)
  * Intermittent pneumatic compression (IPC)
  * 2 h/session, 2× daily, 30-45 mmHg while in bed, continued until independent walking
  * D-dimer blood checks on post-op days 1, 3, 7 and 14; any rise ≥ 20 % or level > 2 mg/L triggers an extra leg ultrasound
  * Continuous safety watch (heart rate, blood pressure, intracranial pressure if monitored); IPC or movement is paused if pressure > 20 mmHg or vital signs become unstable
  All steps are recorded in the electronic nursing chart and coordinated by a neurosurgery-rehabilitation-data
  Interventions: Behavioral: nurse-led program (early movement, leg-sleeve squeezes, and blood tests)
- Standard post-neurosurgical care group (No Intervention): Participants in the control arm receive the hospital's standard post-neurosurgical care, which follows current Chinese and U.S. VTE-guidelines and includes:
  * Routine hydration and general health-education advice
  * Graduated compression stockings (class II, knee-high) worn 8-12 h each day until the patient is walking independently
  * Gentle passive leg movements (about 10 min, 1-2 times daily) when nursing staff judge it safe
  * Low-molecular-weight heparin (40 mg enoxaparin subcutaneous once daily) only for patients judged to be at low bleeding risk (Caprini 4-7) and with no intracranial hemorrhage
  No systematic Caprini re-assessments, no scheduled early-mobilization protocol, no IPC machines, no D-dimer surveillance, and no activity trackers are used.

INTERVENTIONS:
Behavioral: nurse-led program (early movement, leg-sleeve squeezes, and blood tests) — Graded early-movement plan starting within 24 h of surgery
  * Unconscious patients: passive leg exercises 10-15 min, 3× daily
  * Conscious patients: assisted leg, sitting and walking sessions escalated daily (target ≥ 40 min total activity, logged automatically by a wrist-band activity tracker) Intermittent pneumatic compression (IPC)
  * 2 h/session, 2× daily, 30-45 mmHg while in bed, continued until independent walking D-dimer blood checks on post-op days 1, 3, 7 and 14; any rise ≥ 20 % or level > 2 mg/L triggers an extra leg ultrasound Continuous safety watch (heart rate, blood pressure, intracranial pressure if monitored); IPC or movement is paused if pressure > 20 mmHg or vital signs become unstable
  Arms: Nurse-led prevention group

SUMMARY:
The goal of this clinical trial is to see if a nurse-led program (early movement, leg-sleeve squeezes, and blood tests) can prevent dangerous leg blood clots in adults who have just had brain or spine surgery.

Main questions it aims to answer:

* Does the program lower the number of clots within 30 days after surgery?
* Is the program safer and more accurate than the usual clot-risk score nurses already use?

Researchers will compare patients who receive the nurse-led program with patients who receive standard hospital care.

Participants will:

* Be randomly assigned to one of the two groups.
* Have regular leg ultrasounds to check for clots.
* Wear a small activity tracker if they are in the nurse-led group.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Any elective or emergency craniotomy, spinal, or other neurosurgical procedure
* Expected post-operative hospital stay ≥ 3 days
* Patient or legally authorized representative willing and able to give written informed consent

Exclusion Criteria

* Pre-operative ultrasound or imaging proven DVT or pulmonary embolism
* Known hereditary bleeding disorder (e.g., hemophilia) or platelet count < 50 × 10⁹/L
* Chronic therapeutic anticoagulation (warfarin, DOAC, heparin) that cannot be safely stopped, or need for full-dose post-op anticoagulation
* Severe liver disease (Child-Pugh class C) or eGFR < 30 mL/min/1.73 m²
* Life-limiting co-morbidity with expected survival < 30 days
* Pregnancy or breastfeeding
* Current participation in another interventional VTE trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1286 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of objectively confirmed lower-extremity deep-vein thrombosis (DVT) | 30 days
  diagnosed by blinded duplex ultrasound using standard non-compressibility or intraluminal thrombus criteria.

SECONDARY OUTCOMES:
Time from surgery to first objectively confirmed DVT (days) | 30 days
  Time from surgery to first objectively confirmed DVT (days)
All-cause mortality within 30 days | 30 days
  All-cause mortality within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol